CLINICAL TRIAL: NCT02312336
Title: A Safety and Feasibility Study of Transcoronary Myocardial Buffering and Cooling During Primary Coronary Angioplasty to Reduce Myocardial Reperfusion Injury in Acute Myocardial Infarction.
Brief Title: A Pilot Study of Transcoronary Myocardial Cooling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/LO/0476
Record Dates: First submitted 2014-09-18; First posted 2014-12-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Acute Myocardial Infarction
Keywords: ST Elevation Myocardial Infarction; Transcoronary Cooling
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Placebo Comparator): Cohort A - Room temperature coronary perfusate
  Interventions: Other: Cohort A - Room temperature coronary perfusate
- Cohort B (Active Comparator): Cohort B - Cooled coronary perfusate
  Interventions: Other: Cohort B - Cooled coronary perfusate

INTERVENTIONS:
Other: Cohort A - Room temperature coronary perfusate — Patients recruited into the study will receive standard PPCI and in addition a transcoronary infusion of Hartmans solution at room temperature (Cohort A). The research intervention is the infusion of room temperature Hartmans solution.
  Arms: Cohort A
Other: Cohort B - Cooled coronary perfusate — Patients recruited into the study will receive standard PPCI and in addition a transcoronary infusion of Hartmans solution cooled at 15 degrees (Cohort B).
  The research intervention is the infusion of Hartmans solution cooled to 15 degrees.
  Arms: Cohort B

SUMMARY:
Patients with heart attacks caused by blocked coronary arteries are usually treated with a technique called primary angioplasty. Although this treatment is very successful it can result in damage to the heart muscle when the artery is opened due to reperfusion injury. Cooling the entire body has been shown to reduce heart muscle damage during heart attacks in some patients but not in others, however it is uncomfortable due to the shivering, expensive and can result in delays in opening the blocked artery. We are investigating a simpler way to cool the heart muscle directly using cooled fluid passed through the catheter without the shortcomings of entire body cooling. This pilot will address safety and feasibility considerations.

DETAILED DESCRIPTION:
The precise mechanisms involved in ischaemia/reperfusion injury is not fully understood but a number of factors are thought to contribute to cardiac dysfunction14, 15. These include : 1. reperfusion arrhythmias; 2. microvascular obstruction or no-reflow phenomenon; 3. myocardial stunning and 4. cardiomyocyte apoptosis. It is estimated that ischaemia/reperfusion injury occurs in > 30% of patients and is associated with reduced myocardial salvage and poor prognosis16-18. Ischaemia/reperfusion injury may account for up to 50% of the final infarct size9.

Deep hypothermia (< 30 °C) has long been used in protecting the heart during coronary artery bypass grafting and heart transplantation. Intermittent antegrade or retrograde infusion of cold cardioplegia appears to reduce myocardial ischaemia and improves outcome19, 20. Deep hypothermia however can cause spontaneous ventricular fibrillation and impaired cardiac function and its application is limited to the unconscious patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 80 years presenting with ischaemic chest pain of <6 hours and STsegment elevation on the ECG of >0.2 mV in 2 contiguous leads.

Exclusion Criteria:

* Patients with cardiac arrest, previous AMI or CABG, known congestive heart failure, endstage kidney disease or hepatic failure, recent stroke, coagulopathy, pregnancy, or cardiogenic shock.
* Patients who are unable or unwilling to provide assent and informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Symptoms of Chest pain and breathlessness using a Visual Analog Scale | Throughout the PPCI Procedure and for One Hour Afterwards
Haemodynamic changes using the blood pressure (mmHg) and heart rate (beats /min) | Throughout the PPCI Procedure and for One Hour Afterwards
ECG changes (ST segment shift in mm) | Throughout the PPCI Procedure and for One Hour Afterwards
Duration and Volume of perfusate infused used (total time-mins and total volume-mls) | Throughout the PPCI Procedure and for One Hour Afterwards
Intracoronary temperature measured with thermistor wire | Throughout the PPCI Procedure only

SECONDARY OUTCOMES:
Biomarker rise (Cardiac troponin) | 24 hours post PCI procedure
Myocardial infarct size measured with MRI Heart Scan | During hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Miles Dalby, MRCP, MD, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Foundation Trust, Uxbridge, Middlesex, United Kingdom